CLINICAL TRIAL: NCT01365416
Title: Genetic Analysis for Personalised Medicine for Morbid Obesity
Brief Title: Personalised Medicine for Morbid Obesity
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: PMMO
Record Dates: First submitted 2011-06-01; First posted 2011-06-03 (Estimated); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Diabetes
Keywords: diabetes; diabetes remission; obesity; bariatric surgery; gene expression; genetic variation; metabolomics; metabonomics; epigenetic variation; mutations
MeSH Terms: conditions — Diabetes Mellitus; Obesity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — SALIVA BLOOD URINE AND FAECES TISSUE (Muscle, Liver, Subcutaneous fat, Visceral fat)
Oversight: Data Monitoring Committee: No

SUMMARY:
The prevalence of morbid obesity (BMI > 40 kg/m2) is increasing rapidly in the UK, but the investigators lack a coherent strategy for detailed assessment and treatment of the individuals affected, who are at high risk of morbidity and early mortality. The investigators already know that more than 1 in 20 severely-obese individuals have a simple genetic cause of their obesity (usually inherited in an autosomal dominant pattern. Bariatric surgery is the most effective treatment for morbid obesity and certain surgeries can result in the remission of type 2 diabetes. However, some patient fail to achieve the weight loss or experience complications and re-operations. The investigators are unable to predict the outcomes of bariatric surgery particularly in relation to type 2 diabetes remission which is crucial for the assessment of risk to benefit balance before wider future applications of the surgery.

The investigators want to investigate the mechanism underlying Type 2 diabetes remission after bariatric surgery by A) examining the effect of Mendelian forms of obesity and diabetes on T2D remission, B) studying changes in expression profiling patterns in insulin-responsive tissues, C) identifying of eQTLs, and of other genetic variations affecting T2D remission and D) studying the role of epigenetic variation in T2D remission.

DETAILED DESCRIPTION:
SUBJECTS and SAMPLES

Obese patients (n=2000) presenting to Obesity, Endocrine and Medical Clinics at Imperial College Healthcare NHS Trust will be recruited at initial presentation to the service. The patients will be included for this study are patients with BMI >28 kg/m2 and aged between 18-65.

Subjects will undergo blood, saliva, urine and faeces sampling. Patients will also be asked to consent for muscle, liver, subcutaneous and visceral fat tissue collected at the time of surgery. If any of the patients have to undergo a re-operation then blood sample, muscle, liver, subcutaneous and visceral fat tissue will need to be collected again.

Collections of samples from other centres ( e.g Gothenburg) may be analysed in a similar way alongside the samples specified here.

METHODS

The investigators will use methods representing the state-of-the-art at the time of the analysis. Current plans are outlined below:

Standard current methods will be used to extract DNA from saliva or blood and all patients will be screened for monogenic obesity and diabetes.

RNA will be extracted from blood and tissues to perform genome-wide expression analysis.

DNA will be used for performing genome-wide targeted SNP genotyping for the identification of eQTLs, and of genetic variations influencing the outcomes of bariatric surgery.

DNA will be extracted from blood and tissues using standard methods to perform epigenetic analyses.

Patients will be asked to bring an early morning urine sample as well as a faeces sample for later metabonomic/ metagenomic analyses.

Blood samples will also be used for measuring C-peptide, fasting glucose and insulin and other biomarkers as they become available. Subject's weight will be taken at each of the follow-up visits. Subjects will also be analysed for a range of phenotypes concerned with obesity and its co-morbidity as well as for psychological and related outcomes.

PROTOCOL

First point of contact (at group information session):

1. Verbal introduction to study
2. Participant information sheet (Appendix 2)
3. Containers for urine and faeces samples will be handed to patients
4. 1 week follow-up telephone contact for consent to proceed onto first study visit

Visit 1: Screening visit (at pre-surgery assessment (part of routine visit)):

1. Further explanation of study and confirmation of understanding
2. Signed consent form (Appendix 3)
3. Family history questionnaires
4. Measurement of height, weight, head circumference, foot and hand size (supported with Photographic documentation)
5. Psychological questionnaires (these are completed by all patients prior to first study visit upon initial referral to obesity service for audit purposes. Consent will be sought to use these during the first study visit)
6. Blood or saliva
7. Routine blood test to measure C-peptide, fasting glucose and insulin
8. Early morning urine and faeces sample

Visit 2 (during actual surgery):

1. Blood, muscle-, liver-, subcutaneous- and visceral fat tissue

Visit 3 (2 days after surgery):

1. Blood
2. Weight

Visit 4 (10 days post-surgery):

1. Blood
2. Weight
3. Urine

Visit 5 (6 months post-surgery):

1. Blood
2. Weight
3. Urine

   Visit 6 (12 months post-surgery - part of routine follow-up visit):

1 Blood 2 Weight 3 Psychological questionnaires

Visit 7 (18 months post -surgery):

1. Early morning urine and faeces sample
2. Weight

QUESTIONNAIRES

Before the 1st study visit and at 12 months post-surgery, subjects will complete the following questionnaires to assess eating behaviour and personality measures:

1. Eating Disorder Examination Questionnaire (EDEQ) - to identify number of binges per 28 days (Fairburn CG, Beglin S Int Jour. Eat Dis 16:363370, 1994) (Appendix 4).
2. Dutch Eating Behaviour Questionnaire (DEBQ) to measure restraint, emotional and external influences on eating behaviour (Wardle J Psychosom Res 31:1619, 1987) (Appendix 5).

4. Three Factor Eating Questionnaire (TFEQ) - to measure restraint, disinhibition and hunger (Stunkard & Messick. J Psychosom Res 29:7183, 1985) (Appendix 6).

8. Barratt Impulsiveness Scale to measure impulsivity which has been linked to overeating (Patton JM et al J Clin Psych 51: 76874, 1995; Yeomans MR et al. Appetite. 50:46976, 2008) (Appendix 7).

9. PANAS - questionnaire measuring positive and negative affect (Watson, Clark & Tellegen. J Pers Soc Psych 54(6): 10631070, 1988) (Appendix 8).

10. Fagerstrom Test for Nicotine Dependence - a questionnaire assessing current smoking behaviour (Heatherton et al. British Journal of Addiction 86: 1119-1127, 1991) (Appendix 9).

11. Impact of Weight on Quality of Life Questionnaire (IWQOLLite) - a questionnaire measuring the change in subjective quality of life after bariatric surgery (Kolotkin et al. Obesity Research 9: 102111, 2001) (Appendix 10).

12. SF-36 - to assess health of individual patients, to evaluate cost-effectiveness of a treatment and to monitor and compare disease burden (McHorney and Ware, 1995) (Appendix 11).

13. Hospital Anxiety and Depression Scale - to indentify psychiatric disorder or depression (Spinhoven et al., 1997) (Appendix 12).

14. AUDIT drug and alcohol questionnaire (to pick up the early signs of hazardous and harmful drinking and identify mild dependence (Saunders et al., 1993) (Appendix 13).

SALIVA SAMPLING

Saliva samples will be collected using Oragene DNA vials. The acquisition of the saliva sample is done accordingly to the manufacturer's instructions. The patient should not eat, drink, smoke or chew gum for 30 minutes before giving the saliva sample. The patient has to spit into the container until the amount of liquid saliva (not bubbles) reaches at least the level shown in the manufacturer's instructions. The member of staff puts the container on a flat surface, screws the cap onto the container and needs to make sure that the cap is closed tightly. The container has to be mixed gently for at least 10 seconds and kept at room temperature.

BLOOD SAMPLING

At study visit 1-7, venous blood samples will be taken. No more than 100 mls of blood will be taken from each participant during the entire study (no more than 15 mls on each visit). Standard methods will be used to obtain DNA, RNA and serum from blood. Plasma levels of glucose, insulin and C-peptide will be measured by immunoassay.

URINE AND FAECES SAMPLING

Urine and faeces will be collected for metabolomic analysis in 10ml and 20ml Sterilin containers by patients. faeces samples will be collected in sterile containers containing 10 mL of phosphate buffered saline (PBS) (containing, per liter, 8 g of NaCl, 0.2 g of KCl, 1.44 g of Na2HPO4, and 0.24 g of KH2PO4 [pH 7.2]) and stored in home freezers until brought to the laboratory where samples were stored at -80°C until further processing.

TISSUE SAMPLING DURING SURGERY

All biopsies will be taken with scissors and/or Harmonic scalpel (ultrasound instrument for dissection). Muscle tissue will be taken from the abdominal wall at a troachar site. Liver tissue will be taken from the edge of the left liver lobe via needle biopsy. Subcutaneous fat tissue can be taken from an incision for a troachar (about 2 g) and visceral fat tissue can be taken from the major omentum at the greater curvature of the stomach. This will be done at the time of the surgery, and again in any patients requiring re-operation. Standard methods will be used to store the tissues and to stabilize and purify DNA and RNA from the tissues for the purpose of our study.

ELIGIBILITY:
Inclusion Criteria:

* BMI >28 kg/m2
* Age between 18-65 years

Exclusion Criteria:

* donation of blood within the last 3 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 2000 obese patients
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2011-12-09 (Actual); Primary Completion 2025-12-29 (Estimated); Study Completion 2025-12-29 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra I Blakemore, Prof, Principal Investigator — Imperial College London
Locations (1):
- Imperial Weight Centre, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Murphy J, Uttamlal T, Schmidtke KA, Vlaev I, Taylor D, Ahmad M, Alsters S, Purkayastha P, Scholtz S, Ramezani R, Ahmed AR, Chahal H, Darzi A, Blakemore AIF. Tracking physical activity using smart phone apps: assessing the ability of a current app and systematically collecting patient recommendations for future development. BMC Med Inform Decis Mak. 2020 Feb 3;20(1):17. doi: 10.1186/s12911-020-1025-3. PMID 32013996